CLINICAL TRIAL: NCT05204706
Title: A Feasibility Randomised Controlled Trial of a Mobile Phone Application for the Primary Prevention of Type 2 Diabetes in Malaysian Women With Gestational Diabetes Mellitus.
Brief Title: The MalaYsian GestatiOnal Diabetes and Prevention of DiabetES Study
Acronym: MyGODDESS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Putra Malaysia (Other)
Collaborators: King's College London (Other); Ministry of Education, Malaysia (Other Government); Ministry of Health, Malaysia (Other Government)
Responsible Party: Principal Investigator, Boon-How Chew, Principal Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NMRR-21-1667-60212
Record Dates: First submitted 2021-10-31; First posted 2022-01-24 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Gestational Diabetes; GDM; Pregnancy-Induced Diabetes
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Active Comparator): Women who meet study inclusion criteria and consent to study participation will be randomised using sealed envelope randomisation and online database for clinical trials to one of two groups in a 1:1 ratio.
  Interventions: Other: MyManis app
- Control arm (No Intervention): Women allocated to the control arm will receive standard care and no digital intervention. This includes self-monitoring blood glucose and lifestyle advice (diet, physical activity, optimal body weight) by a multidisciplinary team.

INTERVENTIONS:
Other: MyManis app — The women will receive a brochure outlining the app features and step guide on how to download the app which will be available in both Bahasa Melayu and English languages. A link to download the app via text message will also be sent to participants for convenience. Once the app has been downloaded, participants will be invited to set up an account. Once completed this will give them full access to the MyManis app. The key component of MyManis app content presented under six main tabs which are homepage, information, diet, exercise, wellbeing and GDM monitoring. The women will be invited to join group peer support through WhatsApp facilitated by a dietitian trained in motivational interviewing. The women will be notified via text message if an update of the app is required. If there's women who have not accessed the app for over a two-week period will be flagged and a notification will be sent via the app to motivate app engagement.
  Arms: Intervention arm

SUMMARY:
Gestational diabetes mellitus (GDM) is an increasingly common condition of pregnancy and is associated with adverse foetal, infant, and maternal outcomes. Over 50% of women with history of GDM will develop type 2 diabetes (T2D) in later life. Asian women experience disproportionate risk of both GDM and T2D compared to women from other ethnic groups. Lifestyle interventions have been proven to be effective in preventing progression to T2DM in high-risk populations. This is a two-arm, parallel feasibility RCT. Sixty Malaysian women with GDM will be randomized to receive the intervention or standard care in the antenatal period to 12 months postpartum. The intervention is a diabetes prevention intervention delivered via a smartphone application developed based on the Information-Motivation-Behavioral Skills (IMB) model of behavior change and group support utilizing motivational interviewing, which will provide women with tailored information and support to encourage weight loss through adapted dietary intake and physical activity. Women in the control arm will receive standard care.

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM) is a global health challenge, with rates increasing around the world. The adverse short and long-term health outcomes of GDM for both mother and their offspring have been well established. In the long-terms women are up to ten times more likely to develop T2D after GDM and approximately 50% of mothers with GDM will develop diabetes within 10 years. Considerable evidence from several landmark studies has shown that healthy lifestyle interventions and behaviour change can delay or even prevent the onset of T2D in high-risk populations. Given women with prior GDM are at high risk of developing T2D earlier in their lifespan than women with normoglycemic pregnancies, intervening early with an effective diabetes prevention intervention offers a unique window of opportunity along the life-course for the prevention of T2D for the mother. Mobile health (mHealth) is a rapidly growing field of public health, defined as the use of mobile phones and other wireless technology to support the achievement of health objectives. Due to the increasing ownership rate of smartphones, significant numbers of mHealth applications 'apps' have been developed. Pregnant and postpartum women are increasingly utilising such technologies as sources of health information and services for pregnancy self-care and infant care.

The overall aim of the RCT is to test the feasibility of undertaking a definitive trial of a diabetes prevention intervention delivered via a smartphone app over 15-months in women with GDM from randomisation in the antenatal period to 12 months postpartum.

Sixty participants will be recruited from three public health clinics within the southern Selangor state of Malaysia. Women will be eligible for recruitment if they meet the following criteria: i) aged above 18 years, ii) diagnosed with GDM defined using fasting blood glucose > 5.1mmol/1 or 2-hour postprandial >7.8mmol/1 which are the standard guidelines for diagnosis of GDM in Malaysia, iii) permanent resident in the state of Selangor, iv) registered in one of the study health clinics v) owning a smartphone (iOS 11 or Android 7), vi) able to speak, read, and understand English and/or Malay. Women will be excluded if they meet any of the following criteria: i) are having a twin pregnancy, ii) have type 1 or 2 diabetes, iii) have severe physical disability that would prevent any increased uptake of physical exercise, iv) have severe mental illness (psychosis, bipolar, substance dependence or active suicidal ideation), v) are currently participating in a weight loss program or diabetes prevention intervention.

Women who meet study inclusion criteria and consent to study participation will be randomised to either the intervention or control arm. The intervention consists of a smartphone app for women with GDM called MyManis (the English meaning of MyManis is 'my sweet (baby)' and a virtual peer support group. The development of the app was guided by the Information-Motivation-Behavioural Skills (IMB) model of behaviour change. The MyManis app aims to provide women with information and support and motivation to act on this information to make lifestyle behaviour changes in diet and physical activity from pregnancy to post-partum. The app is available for women in both Malay and English. Women allocated to the control arm will receive standard care and no digital intervention.

The overall aim of the RCT is to test the feasibility of undertaking a definitive trial of a diabetes prevention intervention including a smartphone app and group support over 15-months in women with GDM from randomization in the antenatal period to 12 months postpartum.

ELIGIBILITY:
Inclusion Criteria:

* aged above 18 years,
* diagnosed with GDM defined using fasting blood glucose > 5.1mmol/1 or 2-hour postprandial >7.8mmol/1 which are the standard guidelines for diagnosis of GDM in Malaysia,
* permanent resident in the state of Selangor,
* registered in one of the study health clinics
* owning a smartphone (iOS 11 or Android 7) with internet connection,
* able to speak, read, and understand English and/or Malay.

Exclusion Criteria:

* are having a twin pregnancy,
* have type 1 or 2 diabetes,
* have severe physical disability that would prevent any increased uptake of physical exercise,
* have severe mental illness (psychosis, bipolar, substance dependence or active suicidal ideation),
* are currently participating in a weight loss program or diabetes prevention intervention.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — only FEMALE.
Enrollment: 60 (Estimated)
Dates: Start 2022-01-24 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Number of women who were randomised to the treatment groups. | Collected antenatally at 30 weeks pregnancy
  The proportion of women who were randomised (numerator) out of those identified from the clinical registers (study population as denominator)
Number of women that take up the intervention | Collected antenatally at 36 weeks pregnancy
  The proportion of women who take up the intervention (numerator) out of those in the intervention arm (denominator)
Number of women that take up the intervention | Collected antenatally at 6 months after delivery.
  The proportion of women who take up the intervention (numerator) out of those in the intervention arm (denominator)
Number of women that take up the intervention | Collected antenatally at 12 months after delivery.
  The proportion of women who take up the intervention (numerator) out of those in the intervention arm (denominator)
Number of women withdrawn or loss to follow up | Collected antenatally at 36 weeks pregnancy
  The proportion of women who are withdrawn or lost to follow-up (numerator) out of those randomised (denominator)
Number of women withdrawn or loss to follow up | Collected antenatally at 3 months after delivery
  The proportion of women who are withdrawn or lost to follow-up (numerator) out of those randomised (denominator)
Number of women withdrawn or loss to follow up | Collected antenatally at 6 months after delivery
  The proportion of women who are withdrawn or lost to follow-up (numerator) out of those randomised (denominator)
Number of women withdrawn or loss to follow up | Collected antenatally at 9 months after delivery
  The proportion of women who are withdrawn or lost to follow-up (numerator) out of those randomised (denominator)
Number of women withdrawn or loss to follow up | Collected antenatally at 12 months after delivery
  The proportion of women who are withdrawn or lost to follow-up (numerator) out of those randomised (denominator)

SECONDARY OUTCOMES:
Number of women consented | Collected antenatally at 24-28 weeks pregnancy
  The proportion of women who give consent for screening eligibility (numerator) out of those identified from clinical registers (denominator)
Number of women randomised | Collected antenatally at 24-28 weeks pregnancy
  The proportion of women who were randomised (numerator) out of those eligible to participate (denominator)
Number of women completed the secondary outcomes | Collected antenatally at 36 weeks pregnancy
  The proportion of those who completed the secondary outcomes at follow-up (numerator) out of those randomised (denominator)
Number of women completed the secondary outcomes | Collected antenatally at 3 months after delivery
  The proportion of those who completed the secondary outcomes at follow-up (numerator) out of those randomised (denominator)
Number of women completed the secondary outcomes | Collected antenatally at 6 months after delivery
  The proportion of those who completed the secondary outcomes at follow-up (numerator) out of those randomised (denominator)
Number of women completed the secondary outcomes | Collected antenatally at 9 months after delivery
  The proportion of those who completed the secondary outcomes at follow-up (numerator) out of those randomised (denominator)
Number of women completed the secondary outcomes | Collected antenatally at 12 months after delivery
  The proportion of those who completed the secondary outcomes at follow-up (numerator) out of those randomised (denominator)
Number of women randomised | Collected antenatally at 30 weeks pregnancy
  The number of women randomised per month overall, and per month per study site.

OTHER OUTCOMES:
Body weight at T0 | Collected antenatally at T0: 30 weeks pregnancy
  Weight (kg)
Body weight at T1 | Collected antenatally at T1: 36 weeks pregnancy
  Weight (kg)
Body weight at T2 | Collected antenatally at T2: 3 months after delivery
  Weight (kg)
Body weight at T3 | Collected antenatally at T3: 6 months after delivery
  Weight (kg)
Body weight at T4 | Collected antenatally at T4: 9 months after delivery
  Weight (kg)
Body weight at T5 | Collected antenatally at T5: 12 months after delivery
  Weight (kg)
Height at T0 | Collected antenatally at T0: 30 weeks pregnancy
  measured for 1 time only (in centimetres, cm)
Body mass index at T0 | Collected antenatally at T0: 30 weeks pregnancy
  calculated as body weight divided by (heightxheight) (kg/m^2)
Body mass index at T1 | Collected antenatally at T1: 36 weeks pregnancy
  calculated as body weight divided by (heightxheight) (kg/m^2)
Body mass index at T2 | Collected antenatally at T2: 3 months after delivery
  calculated as body weight divided by (heightxheight) (kg/m^2)
Body mass index at T3 | Collected antenatally at T3: 6 months after delivery
  calculated as body weight divided by (heightxheight) (kg/m^2)
Body mass index at T4 | Collected antenatally at T4: 9 months after delivery
  calculated as body weight divided by (heightxheight) (kg/m^2)
Body mass index at T5 | Collected antenatally at T5: 12 months after delivery
  calculated as body weight divided by (heightxheight) (kg/m^2)
Body fat percentage at T0 | Collected antenatally at T0: 30 weeks pregnancy
  Body fat percentage reported in % (to 1 decimal point)
Body fat percentage at T1 | Collected antenatally at T1: 36 weeks pregnancy
  Body fat percentage reported in % (to 1 decimal point)
Body fat percentage at T2 | Collected antenatally at T2: 3 months after delivery
  Body fat percentage reported in % (to 1 decimal point)
Body fat percentage at T3 | Collected antenatally at T3: 6 months after delivery
  Body fat percentage reported in % (to 1 decimal point)
Body fat percentage at T4 | Collected antenatally at T4: 9 months after delivery
  Body fat percentage reported in % (to 1 decimal point)
Body fat percentage at T5 | Collected antenatally at T5: 12 months after delivery
  Body fat percentage reported in % (to 1 decimal point)
Blood pressure reading at T0 | Collected antenatally at T0: 30 weeks pregnancy
  measure systolic and diastolic blood pressure (mmHg)
Blood pressure reading at T1 | Collected antenatally at T1: 36 weeks pregnancy
  measure systolic and diastolic blood pressure (mmHg)
Blood pressure reading at T3 | Collected antenatally at T3: 6 months after delivery
  measure systolic and diastolic blood pressure (mmHg)
Blood pressure reading at T5 | Collected antenatally at T5: 12 months after delivery
  measure systolic and diastolic blood pressure (mmHg)
Total Cholestrol at T0 | Collected antenatally at T0: 30 weeks pregnancy
  Total Cholestrol (mmol/L)
Total Cholestrol at T1 | Collected antenatally at T1: 36 weeks pregnancy
  Total Cholestrol (mmol/L)
Total Cholestrol at T3 | Collected antenatally at T3: 6 months after delivery
  Total Cholestrol (mmol/L)
Total Cholestrol at T5 | Collected antenatally at T5: 12 months after delivery
  Total Cholestrol (mmol/L)
Low Density Lipoprotein Cholestrol at T0 | Collected antenatally at T0: 30 weeks pregnancy
  Low Density Lipoprotein Cholestrol, LDL (mmol/L)
Low Density Lipoprotein Cholestrol at T1 | Collected antenatally at T1: 36 weeks pregnancy
  Low Density Lipoprotein Cholestrol, LDL (mmol/L)
Low Density Lipoprotein Cholestrol at T3 | Collected antenatally at T3: 6 months after delivery
  Low Density Lipoprotein Cholestrol, LDL (mmol/L)
Low Density Lipoprotein Cholestrol at T5 | Collected antenatally at T5: 12 months after delivery
  Low Density Lipoprotein Cholestrol, LDL (mmol/L)
High Density Lipoprotein cholesterol at T0 | Collected antenatally at T0: 30 weeks pregnancy
  High Density Lipoprotein cholesterol, HDL (mmol/L)
High Density Lipoprotein cholesterol at T1 | Collected antenatally at T1: 36 weeks pregnancy
  High Density Lipoprotein cholesterol, HDL (mmol/L)
High Density Lipoprotein cholesterol at T3 | Collected antenatally at T3: 6 months after delivery
  High Density Lipoprotein cholesterol, HDL (mmol/L)
High Density Lipoprotein cholesterol at T5 | Collected antenatally at T5: 12 months after delivery
  High Density Lipoprotein cholesterol, HDL (mmol/L)
HbA1c at T0 | Collected antenatally at T0: 30 weeks pregnancy
  HbA1c (%)
HbA1c at T1 | Collected antenatally at T1: 36 weeks pregnancy
  HbA1c (%)
HbA1c at T3 | Collected antenatally at T3: 6 months after delivery
  HbA1c (%)
HbA1c at T5 | Collected antenatally at T5: 12 months after delivery
  HbA1c (%)
Fasting blood glucose at T0 | Collected antenatally at T0: 30 weeks pregnancy
  Fasting blood glucose (mmol/l)
Fasting blood glucose at T1 | Collected antenatally at T1: 36 weeks pregnancy
  Fasting blood glucose (mmol/l)
Oral glucose tolerance test (OGTT) Fasting at T3 | Collected antenatally at T3: 6 months after delivery
  Oral glucose tolerance test (OGTT) Fasting (mmol/l)
Oral glucose tolerance test (OGTT) Fasting at T5 | Collected antenatally at T5: 12 months after delivery
  Oral glucose tolerance test (OGTT) Fasting (mmol/l)
Oral glucose tolerance test (OGTT) 2-hour Postprandial at T3 | Collected antenatally at T3: 6 months after delivery
  Oral glucose tolerance test (OGTT) 2-hour Postprandial (mmol/l)
Oral glucose tolerance test (OGTT) 2-hour Postprandial at T5 | Collected antenatally at T5: 12 months after delivery
  Oral glucose tolerance test (OGTT) 2-hour Postprandial (mmol/l)
Fasting Serum Insulin at T0 | Collected antenatally at T0: 30 weeks pregnancy
  Fasting Serum Insulin (U/mL)
Fasting Serum Insulin at T1 | Collected antenatally at T1: 36 weeks pregnancy
  Fasting Serum Insulin (U/mL)
Fasting Serum Insulin at T3 | Collected antenatally at T3: 6 months after delivery
  Fasting Serum Insulin (U/mL)
Fasting Serum Insulin at T5 | Collected antenatally at T5: 12 months after delivery
  Fasting Serum Insulin (U/mL)
Insulin resistance at T0 | Collected antenatally at T0: 30 weeks pregnancy
  Insulin resistance (HOMA-IR)
Insulin resistance at T1 | Collected antenatally at T1: 36 weeks pregnancy
  Insulin resistance (HOMA-IR)
Insulin resistance at T3 | Collected antenatally at T3: 6 months after delivery
  Insulin resistance (HOMA-IR)
Insulin resistance at T5 | Collected antenatally at T5: 12 months after delivery
  Insulin resistance (HOMA-IR)
Total score for Self-efficacy for exercise at T0 | Collected at T0: 30 weeks pregnancy
  This scale consist of 18 items whereby the response options are ranging from 0-100, ranging in 10-unit intervals from 0 (cannot do); through intermediate degrees of assurance, 50 (moderately certain can do); to complete assurance, 100 (highly certain can do). The scale is scored by summing the numerical ratings for each response and dividing by the number of responses. Higher scores indicates higher self-efficacy for exercise.
Total score for Self-efficacy for exercise at T3 | Collected at T3: 6 months after delivery
  This scale consist of 18 items whereby the response options are ranging from 0-100, ranging in 10-unit intervals from 0 (cannot do); through intermediate degrees of assurance, 50 (moderately certain can do); to complete assurance, 100 (highly certain can do). The scale is scored by summing the numerical ratings for each response and dividing by the number of responses. Higher scores indicates higher self-efficacy for exercise.
Total score for Self-efficacy for exercise at T5 | Collected at T5: 12 months after delivery
  This scale consist of 18 items whereby the response options are ranging from 0-100, ranging in 10-unit intervals from 0 (cannot do); through intermediate degrees of assurance, 50 (moderately certain can do); to complete assurance, 100 (highly certain can do). The scale is scored by summing the numerical ratings for each response and dividing by the number of responses. Higher scores indicates higher self-efficacy for exercise.
Mother-infant relationship at T0 | Collected at 30 weeks pregnancy
  The mother-infant relationship will be assessed using the Maternal Antenatal Attachment Scale which comprises 19 items with response options presented on a 5-point Likert scale. A total score is obtained by summing the responses to the 19 items, resulting in a possible scoring range of 19 to 95. Higher scores are indicative of stronger attachment.
Mother-infant relationship at T3 | Collected at 6 months after delivery
  The mother-infant relationship will be assessed using the Maternal Antenatal Attachment Scale which comprises 19 items with response options presented on a 5-point Likert scale. A total score is obtained by summing the responses to the 19 items, resulting in a possible scoring range of 19 to 95. Higher scores are indicative of stronger attachment.
Mother-infant relationship at T5 | Collected at 12 months after delivery
  The mother-infant relationship will be assessed using the Maternal Antenatal Attachment Scale which comprises 19 items with response options presented on a 5-point Likert scale. A total score is obtained by summing the responses to the 19 items, resulting in a possible scoring range of 19 to 95. Higher scores are indicative of stronger attachment.
Depressive symptoms at T0 | Collected at T0: 30 weeks pregnancy
  The questionnaire consist of 10 items. Add up all checked (Tick) boxes on PHQ-9. For every tick boxes: the score indicated is as below: 0= Not at all; 1=Several days; 2=More than half the days; 3=Nearly every day. Then add the subtotal to produce a total score. The possible range score is 0-27.
Depressive symptoms at T3 | Collected at T3: 6 months after delivery
  The questionnaire consist of 10 items. Add up all checked (Tick) boxes on PHQ-9. For every tick boxes: the score indicated is as below: 0= Not at all; 1=Several days; 2=More than half the days; 3=Nearly every day. Then add the subtotal to produce a total score. The possible range score is 0-27.
Depressive symptoms at T5 | Collected at T5: 12 months after delivery
  The questionnaire consist of 10 items. Add up all checked (Tick) boxes on PHQ-9. For every tick boxes: the score indicated is as below: 0= Not at all; 1=Several days; 2=More than half the days; 3=Nearly every day. Then add the subtotal to produce a total score. The possible range score is 0-27.
Dietary intake at T0 | Collected at T0: 30 weeks pregnancy
  Total macronutrient intake from standardised multiple-pass 24-hour dietary recall)
Dietary intake at T3 | Collected at T3: 6 months after delivery
  Total macronutrient intake from standardised multiple-pass 24-hour dietary recall)
Dietary intake at T5 | Collected at T5: 12 months after delivery
  Total macronutrient intake from standardised multiple-pass 24-hour dietary recall)
Physical activity at T0 | Collected at T0: 30 weeks pregnancy
  The questionnaire consist of 7 items. The total score will be reported as a continuous measure and reported as median METminutes. Median values can be computed for walking (W), moderate-intensity activities (M), and vigorous-intensity activities (V) using the following formulas:
  MET values and Formula for computation of Met-minutes Walking MET-minutes/week = 3.3 * walking minutes * walking days Moderate MET-minutes/week = 4.0 * moderate-intensity activity minutes * moderate days Vigorous MET-minutes/week = 8.0 * vigorous-intensity activity minutes * vigorous-intensity days A combined total physical activity MET-min/week can be computed as the sum of Walking + Moderate + Vigorous MET-min/week scores.
Physical activity at T3 | Collected at T3: 6 months after delivery
  The questionnaire consist of 7 items. The total score will be reported as a continuous measure and reported as median METminutes. Median values can be computed for walking (W), moderate-intensity activities (M), and vigorous-intensity activities (V) using the following formulas:
  MET values and Formula for computation of Met-minutes Walking MET-minutes/week = 3.3 * walking minutes * walking days Moderate MET-minutes/week = 4.0 * moderate-intensity activity minutes * moderate days Vigorous MET-minutes/week = 8.0 * vigorous-intensity activity minutes * vigorous-intensity days A combined total physical activity MET-min/week can be computed as the sum of Walking + Moderate + Vigorous MET-min/week scores.
Physical activity at T5 | Collected at T5: 12 months after delivery
  The questionnaire consist of 7 items. The total score will be reported as a continuous measure and reported as median METminutes. Median values can be computed for walking (W), moderate-intensity activities (M), and vigorous-intensity activities (V) using the following formulas:
  MET values and Formula for computation of Met-minutes Walking MET-minutes/week = 3.3 * walking minutes * walking days Moderate MET-minutes/week = 4.0 * moderate-intensity activity minutes * moderate days Vigorous MET-minutes/week = 8.0 * vigorous-intensity activity minutes * vigorous-intensity days A combined total physical activity MET-min/week can be computed as the sum of Walking + Moderate + Vigorous MET-min/week scores.
mean step count at T0 | Collected at T0: 30 weeks pregnancy
  Number of steps in inbuild smartphone app
mean step count at T3 | Collected at T3: 6 months after delivery
  Number of steps in inbuild smartphone app
mean step count at T5 | Collected at T5: 12 months after delivery
  Number of steps in inbuild smartphone app
Infant feeding T3 | Collected at T3: 6 months after delivery
  Type of feeding status
Infant feeding at T5 | Collected at T5: 12 months after delivery
  Type of feeding status
Alcohol intake at T0 | Collected at T0: 30 weeks pregnancy
  Frequency of intake
Alcohol intake at T3 | Collected at T3: 6 months after delivery
  Frequency of intake
Alcohol intake at T5 | Collected at T5: 12 months after delivery
  Frequency of intake
Smoking status at T0 | Collected at T0: 30 weeks pregnancy
  type of smoker
Smoking status at T3 | Collected at T3: 6 months after delivery
  type of smoker
Smoking status at T5 | Collected at T5: 12 months after delivery
  type of smoker
Recruitment rate | Collected at 30 weeks pregnancy
  number of eligible, consented, screened, enrolled, and randomised
T1 Dosage delivered - app download | Collected at T1: 36 weeks pregnancy
  The number of MyManis app delivered by the researcher and the number of app downloads (n) by the participant.
T3 Dosage delivered - app download | Collected at T3: 6 months after delivery
  The number of MyManis app delivered by the researcher and the number of app downloads (n) by the participant.
T5 Dosage delivered - app download | Collected at T5: 12 months after delivery
  The number of MyManis app delivered by the researcher and the number of app downloads (n) by the participant.
T1 Dosage delivered - Support group | Collected at T1: 36 weeks pregnancy
  Total number of group support sessions (n) planned to deliver by the dietitian train in motivational interviewing.
T3 Dosage delivered - Support group | Collected at T3: 6 months after delivery
  Total number of group support sessions (n) planned to deliver by the dietitian train in motivational interviewing.
T5 Dosage delivered - Support group | Collected at T5: 12 months after delivery
  Total number of group support sessions (n) planned to deliver by the dietitian train in motivational interviewing.
T1 Dosage received - Participant's engagement | Collected at T1: 36 weeks pregnancy
  The number of participant log into MyManis app per month (n)
T3 Dosage received - Participant's engagement | Collected at T3: 6 months after delivery
  The number of participant log into MyManis app per month (n)
T5 Dosage received - Participant's engagement | Collected at T5: 12 months after delivery
  The number of participant log into MyManis app per month (n)
T1 Dosage received - length of log in | Collected at T1: 36 weeks pregnancy
  This is an extent to which participant's engagement through length of participant log into MyManis app (hours and minutes)
T3 Dosage received - length of log in | Collected at T3: 6 months after delivery
  This is an extent to which participant's engagement through length of participant log into MyManis app (hours and minutes)
T5 Dosage received - length of log in | Collected at T5: 12 months after delivery
  This is an extent to which participant's engagement through length of participant log into MyManis app (hours and minutes)
T1 Dosage received - time spent on DIET component | Collected at T1: 36 weeks pregnancy
  Participant time spent on DIET component (hours and minutes)
T1 Dosage received - time spent on EXERCISE component | Collected at T1: 36 weeks pregnancy
  Participant time spent on EXERCISE component (hours and minutes)
T1 Dosage received - time spent on MENTAL HEALTH component | Collected at T1: 36 weeks pregnancy
  Participant time spent on MENTAL HEALTH component (hours and minutes)
T3 Dosage received - time spent on DIET component | Collected at T3: 6months after delivery
  Time spent on DIET component (hours and minutes)
T3 Dosage received - time spent on EXERCISE component | Collected at T3: 6months after delivery
  Time spent on EXERCISE component (hours and minutes)
T3 Dosage received - time spent on MENTAL HEALTH component | Collected at T3: 6months after delivery
  Time spent on MENTAL HEALTH component (hours and minutes)
T5 Dosage received - time spent on DIET component | Collected at T5: 12 months after delivery
  Time spent on DIET component (hours and minutes)
T5 Dosage received - time spent on EXERCISE component | Collected at T5: 12 months after delivery
  Time spent on EXERCISE component (hours and minutes)
T5 Dosage received - time spent on MENTAL HEALTH component | Collected at T5: 12 months after delivery
  Time spent on MENTAL HEALTH component (hours and minutes)
Fidelity at T1 | collected at T1: 36 weeks pregnancy
  This is an assessment of the researcher in the team to check on the research dietitian's in delivering group support according to a pre-specified plan. This will be reported descriptively.
Fidelity at T3 | collected at T3: 6 months after delivery
  This is an assessment of the researcher in the team to check on the research dietitian's in delivering group support according to a pre-specified plan. This will be reported descriptively.
Fidelity at T5 | collected at T5: 12 months after delivery
  This is an assessment of the researcher in the team to check on the research dietitian's in delivering group support according to a pre-specified plan. This will be reported descriptively.
Semi-structured interview at T1 | Collected at T1: 36 weeks pregnancy
  Interviews on participant experiences and satisfaction towards the intervention
Semi-structured interview at T3 | Collected at T3: 6 months after delivery
  Interviews on participant experiences and satisfaction towards the intervention
Semi-structured interview at T5 | Collected at T5: 12 months after delivery
  Interviews on participant experiences and satisfaction towards the intervention
Mother infant relationship at T2 | Collected at T2: 3 months after delivery
  3-minutes video recording captured through Zoom and coded based on the CARE-INDEX
Satisfaction survey at T5 | Collected at T5: 12 months after delivery
  acceptability, experience and perceived usefulness of the project
Hypertension | Collected at T2: 3 months postpartum
  This is a diagnosis by the clinic and reported in the record from anytime after delivery to 3 months postpartum.
Hypercholesterolemia | Collected at T2: 3 months postpartum
  This is a diagnosis by the clinic and reported in the record from anytime after delivery to 3 months postpartum.
Delivery method | Collected at T2: 3 months postpartum
  This is reported in the record from anytime after delivery to 3 months postpartum.
Pregnancy complications | Collected at T2: 3 months postpartum
  This is reported in the record from anytime after delivery to 3 months postpartum.
Birth complications | Collected at T2: 3 months postpartum
  This is reported in the record from anytime after delivery to 3 months postpartum.
Breastfeeding status on discharge | Collected at T2: 3 months postpartum
  This is reported in the record from anytime after delivery to 3 months postpartum.
Neonatal birth weight | Collected at T2: 3 months postpartum
  This is reported in the record from anytime after delivery to 3 months postpartum.
Neonatal APGAR score 5 minutes | Collected at T2: 3 months postpartum
  This is reported in the record from anytime after delivery to 3 months postpartum.
Congenital anomaly | Collected at T2: 3 months postpartum
  This is reported in the record from anytime after delivery to 3 months postpartum.
Congenital pnuemonia / heart defects | Collected at T2: 3 months postpartum
  This is reported in the record from anytime after delivery to 3 months postpartum.
Admission to neonatal intensive care | Collected at T2: 3 months postpartum
  This is reported in the record from anytime after delivery to 3 months postpartum.
Length of stay at the hospital ward | Collected at T2: 3 months postpartum
  This is reported in the record from anytime after delivery to 3 months postpartum.

CONTACTS AND LOCATIONS:
Overall Officials: BOON HOW CHEW, Principal Investigator — Universiti Putra Malaysia; KHALIDA ISMAIL, Principal Investigator — King's College London
Locations (3):
- Malaysia (3):
  - Klinik Kesihatan Putrajaya Presint 9, Putrajaya, Kuala Lumpur
  - Klinik Kesihatan Puchong Batu 14, Petaling Jaya, Selangor
  - Klinik Kesihatan Seri Kembangan, Seri Kembangan, Selangor

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mohd Sa'id, I. I., Papachristou Nadal, I., Forbes, A., Goldsmith, K., Ismail, I. Z., Hassan, F., Ching, S. M., Guess, N., Murphy, H., Prina, M., Mohd Yusoff, B. N., Basri, N. I., Binti Salim, M. S., Mahamad Sobri, N. H., Har Yap, P. P., Ismail, K., & Chew, B. H. (2021). A Protocol of Process Evaluations of Interventions for the Prevention of Type 2 Diabetes in Women With Gestational Diabetes Mellitus: A Systematic Review. International Journal of Qualitative Methods, 20. https://doi.org/10.1177/16094069211034010
- [Background] Sobri NHM, Ismail IZ, Hassan F, Papachristou Nadal I, Forbes A, Ching SM, Ali H, Goldsmith K, Murphy H, Guess N, Mohd Yusof BN, Basri NI, Salim MS, Azmiyaty C, Mohd Sa'id II, Chew BH, Ismail K; MYGODDESS Project Team. Protocol for a qualitative study exploring the perception of need, importance and acceptability of a digital diabetes prevention intervention for women with gestational diabetes mellitus during and after pregnancy in Malaysia (Explore-MYGODDESS). BMJ Open. 2021 Aug 26;11(8):e044878. doi: 10.1136/bmjopen-2020-044878. PMID 34446477
- [Background] Benton M, Iman I, Goldsmith K, Forbes A, Ching SM, Papachristou Nadal I, Guess N, Murphy HR, Mohd Yusof BN, Baharom A, Mahamad Sobri NH, Basri NI, Salim MS, Ismail IZ, Hassan F, Ismail K, Chew BH. A Mobile Phone App for the Prevention of Type 2 Diabetes in Malaysian Women With Gestational Diabetes Mellitus: Protocol for a Feasibility Randomized Controlled Trial. JMIR Res Protoc. 2022 Sep 8;11(9):e37288. doi: 10.2196/37288. PMID 36074545
- See also: UKRI website about the project — https://gtr.ukri.org/projects?ref=MR%2FT018240%2F1